CLINICAL TRIAL: NCT05158881
Title: Use of Near-infrared Spectroscopy in Cerebral Oxygenation Monitoring in Full Term Neonates During Transition After Birth
Brief Title: Near-infrared Spectroscopy in Cerebral Oxygenation Monitoring in Full Term Neonates
Status: Completed | Type: Observational
Sponsor: Marwa Mohamed Farag (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Farag, Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: 0106540
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Cerebral Oxygenation in Full-term Neonates
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonates delivered by normal vaginal delivery
  Interventions: Device: Near-infrared spectroscopy
- Neonates delivered by elective cesarean section.
  Interventions: Device: Near-infrared spectroscopy

INTERVENTIONS:
Device: Near-infrared spectroscopy — Near-infrared spectroscopy (NIRS) offers the non-invasive continuous monitoring of cerebral oxygenation and perfusion. Cerebral regional oxygen (crSO2) measured via NIRS represents a mixed tissue saturation value, thus enabling information on the balance of cerebral oxygen delivery and oxygen consumption.

SUMMARY:
The aim of the study was to assess the values of cerebral oxygenation in full-term neonates in the first 10 minutes of life and to compare these values between neonates delivered by normal vaginal delivery and those delivered by elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥38 weeks, without any medical support and normal pregnancy development.

Exclusion Criteria:

* Newborns with gestational age <38 weeks.
* Newborns with intrauterine growth restriction.
* Evidence of perinatal depression (hypoxic ischemic encephalopathy).
* The need for respiratory support or oxygen therapy in the first 10 minutes of life.
* Suspected or known brain malformations or congenital cyanotic heart disease.
* Birth complications (e.g. vacuum extraction or forceps application).
* Newborn delivered through cesarean section with previous attempts of normal vaginal delivery.

Ages: 0 Minutes to 10 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full term neonates born either via normal vaginal delivery or elective cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Cerebral regional oxygen saturation monitoring (crSO2) | the first 10 minutes of life
  Measurements was done by using Near infrared spectroscopy (INVOSTM 5100C Cerebral/ Somatic Oximeter Monitor; Covidien) by placing a neonatal brain sensor on the left frontoparietal area of the newborn's head.
Peripheral oxygen saturation monitoring (SpO2) | the first 10 minutes of life
  Oxygen saturation was measured using pulse oximeter (Masimo or Nellcor) by applying a preductal pulseoximetry sensor to the right wrist.
Blood gas analysis | up to 10 minutes of life
  It was performed from umbilical cord blood. All newborns will be clinically observed and evaluated during this period by a neonatologist, and clinical status will be assessed by Apgar score. The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Fractional tissue oxygen extraction (FTOE) | up to 10 minutes of life
  After measuring peripheral oxygen saturation (SpO2) and cerebral regional oxygen saturation (crSO2).
  For evaluation of the balance of oxygen delivery and oxygen consumption, calculation of the fractional tissue oxygen extraction can be done using the following equation:
  FTOE=(SpO2-crSO2)/SpO2

CONTACTS AND LOCATIONS:
Overall Officials: Alaa IA Ibrahim, MBBCh, Principal Investigator — Faculty of Medicine, Alexandria University, Egypt; Hesham A Ghazal, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt; Marwa M Farag, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt; Bahaa S Hammad, Study Director — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt